CLINICAL TRIAL: NCT03791580
Title: Reducing High-Risk Geriatric Polypharmacy Via EHR Nudges: Pilot Phase
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: NIA funded the first phase of the R21. The clinical trial never began as the R33 was not supported.
Sponsor: RAND (Other)
Collaborators: Northwestern University (Other); University of California, Los Angeles (Other); University of Southern California (Other); University of Pittsburgh (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: STU00207210; R21AG057396 (NIH)
Record Dates: First submitted 2018-12-29; First posted 2019-01-02 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Fall; Congestive Heart Failure; Chronic Kidney Failure; Adverse Drug Event
Keywords: Polypharmacy; Primary Health Care; Economics, Behavioral; Deprescriptions; Decision Support Systems, Clinical; Electronic Health Records; Geriatrics
MeSH Terms: conditions — Heart Failure; Kidney Failure, Chronic; Drug-Related Side Effects and Adverse Reactions; Behavior

STUDY DESIGN:
Intervention Model Description: The investigators will randomly assign each of the 3 participating pilot practices to 1 of 3 arms: (1) commitment nudge, (2) justification nudge, or (3) both commitment and justification nudges. Randomization will be at the practice level, without replacement, thus assigning exactly 1 practice to each arm. All participating clinicians within a given practice will receive the same nudges. Northwestern-affiliated practices that do not participate in the pilot will constitute a fourth arm of this pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Commitment nudge (Experimental): Primary care clinicians in the practice assigned to this arm will receive only the commitment nudge.
  Interventions: Behavioral: Commitment nudge
- Justification nudge (Experimental): Primary care clinicians in the practice assigned to this arm will receive only the justification nudge.
  Interventions: Behavioral: Justification nudge
- Commitment + Justification nudges (Experimental): Primary care clinicians in the practice assigned to this arm will receive both the commitment nudge and the justification nudge.
  Interventions: Behavioral: Commitment nudge; Behavioral: Justification nudge
- Non-participating (No Intervention): Primary care clinicians in Northwestern-affiliated practices other than the 3 pilot-participating practices will not receive any study interventions.

INTERVENTIONS:
Behavioral: Commitment nudge — The commitment nudge will ask clinicians to commit to discussing high-risk polypharmacy at the next office visit with patients who have high-risk polypharmacy. Clinicians who commit will receive a reminder just before the next office visit begins. The patient will also receive notification of the commitment via EHR patient portal.
  This nudge will be operationalized via two sequential clinician-facing EHR best practice alerts (BPAs): the first at time of opening any encounter (including encounters other than a face-to-face office visit, e.g., medication refills), and the second (contingent on making a commitment to discuss high-risk polypharmacy) at time of opening the subsequent encounter for a face-to-face office visit. Each of these BPAs will describe the specific high-risk polypharmacy criterion (or criteria) the patient meets, the specific harms associated with the medication(s) triggering the criterion/criteria, and lower-risk alternative treatment strategies.
  Arms: Commitment + Justification nudges; Commitment nudge
Behavioral: Justification nudge — The justification nudge will ask clinicians who prescribe or renew a drug that meets high-risk polypharmacy criteria (in the context of the patient's other medications) to write a brief justification for prescribing this high-risk medication. This written justification will be recorded in the patient's medical record. The best practice alert requesting the justification will also describe the specific high-risk polypharmacy criterion (or criteria) the patient meets, the specific harms associated with the medication(s) triggering the criterion/criteria, and lower-risk alternative treatment strategies.
  Arms: Commitment + Justification nudges; Justification nudge

SUMMARY:
Polypharmacy is common among older adults in the United States and is associated with harms such as adverse drug reactions and higher costs of care. This pilot-phase project is designed to test two electronic health record (EHR)-based behavioral economic nudges to help primary care clinicians reduce the rate of high-risk polypharmacy among their older adult patients.

DETAILED DESCRIPTION:
Polypharmacy increases the likelihood of being prescribed and harmed by high-risk medications. As noted in the 2014 National Action Plan for Adverse Drug Event (ADE) Prevention, polypharmacy both increases the likelihood of being prescribed high-risk medications and increases the likelihood that these high-risk medications will lead to adverse drug events. This pilot-phase study is intended to test clinicians' perceptions of EHR-based nudges designed to reduce high-risk polypharmacy among patients aged 65 years or more, thereby enabling investigators to refine the nudges, and to generate outcomes data that will inform power calculations for a subsequent larger study (the main study) of the nudges' effectiveness.

In this pilot-phase study, the investigators will deploy 2 EHR-based behavioral nudges (a commitment nudge and a justification nudge) among 18 or more primary care clinicians in 3 primary care practices (6 clinicians or more per practice) affiliated with Northwestern University for approximately 4 months. The 3 practices participating in the pilot will be a convenience sample of Northwestern-affiliated practices known to study investigators.

The investigators will randomly assign each of the 3 participating pilot practices to 1 of 3 arms: (1) commitment nudge, (2) justification nudge, or (3) both commitment and justification nudges. Randomization will be at the practice level, without replacement, thus assigning exactly 1 practice to each arm. All participating clinicians within a given practice will receive the same nudges.

Northwestern-affiliated practices that do not participate in the pilot will constitute a fourth arm of this pilot study.

The investigators will ask leaders of participating practices for their qualitative observations on how clinicians and patients experience the nudges (e.g., how the nudges affect workflows). The investigators also will collect data on the outcome measures before and during the approximately 4-month pilot period and compare these data to contemporaneous outcomes measures generated by Northwestern-affiliated practices that do not participate in the pilot.

ELIGIBILITY:
Inclusion Criteria:

* Primary care clinicians practicing in one of the participating Northwestern-affiliated practices

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
High-risk polypharmacy criterion: Fall condition-drug interaction | 28 months
  Denominator: count of patients aged >=65 years AND who have >=1 fall marker within the prior 2 years (ICD-10 codes for falls or hip fractures; OR who are recorded in the EHR as being high-risk for falls). Numerator: count of patients in the denominator who have 5+ medications in their EHR med list AND who have >=1 medication in their EHR med list that is a tricyclic antidepressant, Z-drug (e.g., zolpidem), benzodiazepine, antipsychotic, anticonvulsant, SSRI/SNRI, or opioid.
High-risk polypharmacy criterion: Fall drug-drug interaction | 28 month
  Denominator: count of patients aged >=65 years. Numerator: count of patients in the denominator who have 5+ meds AND who have >=3 medications in their EHR med list that are tricyclic antidepressants, Z-drugs (e.g., zolpidem), benzodiazepines, antipsychotics, anticonvulsants, SSRIs/SNRIs, or opioids.
High-risk polypharmacy criterion: CKD-glyburide/glimepiride interaction | 28 months
  Denominator: count of patients aged >=65 years AND who have most-recent estimated glomerular filtration rate (eGFR) < 60 as estimated by the Cockcroft-Gault equation. Numerator: count of patients in the denominator who have 5+ meds AND glyburide or glimepiride in their EHR med list.
High-risk polypharmacy criterion: CKD-NSAID interaction | 28 months
  Denominator: count of patients aged >=65 years AND who have most-recent eGFR < 30 as estimated by the Cockcroft-Gault equation. Numerator: count of patients in the denominator who have 5+ meds AND a systemically-absorbed non-steroidal anti-inflammatory drug (NSAID) in their EHR med list.
High-risk polypharmacy criterion: CHF-NSAID interaction | 28 months
  Denominator: count of patients aged >=65 years AND who have 5+ meds AND congestive heart failure (identified via ICD-10 code within prior 2 years). Numerator: count of patients in the denominator who have a systemically-absorbed non-steroidal anti-inflammatory drug (NSAID) in their EHR med list.
High-risk polypharmacy criterion: CHF-non-dihydropyridine calcium channel blocker interaction | 28 months
  Denominator: count of patients aged >=65 years AND who have low-ejection-fraction congestive heart failure (identified via ICD-10 code within prior 2 years). Numerator: count of patients in the denominator who have 5+ meds AND a non-dihydropyridine calcium channel blocker in their EHR med list.
High-risk polypharmacy criterion: CHF-thiazolidinedione interaction | 28 months
  Denominator: count of patients aged >=65 years AND who have low-ejection-fraction congestive heart failure (identified via ICD-10 code within prior 2 years). Numerator: count of patients in the denominator who have 5+ meds AND a thiazolidinedione in their EHR med list.

CONTACTS AND LOCATIONS:
Overall Officials: Mark W Friedberg, MD, MPP, Principal Investigator — RAND
Locations (1):
- Northwestern Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No